CLINICAL TRIAL: NCT06114082
Title: Transarterial Chemoembolization Using Idarubicin Versus Doxorubicin Chemoemulsion in Patients with Hepatocellular Carcinoma (IDADOX)
Brief Title: TACE Using Idarubicin Versus Doxorubicin Chemoemulsion in Patients with Hepatocellular Carcinoma
Acronym: IDADOX
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Guerbet (Industry)
Responsible Party: Principal Investigator, Jin Woo Choi, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-2211-153-1381
Record Dates: First submitted 2023-10-19; First posted 2023-11-02 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer
Keywords: Hepatocellular carcinoma; Transarterial chemoembolization; Doxorubicin; Idarubicin
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IDA-TACE (Experimental): Patients treated by conventional TACE using idarubicin chemoemulsion
  Interventions: Procedure: IDA-TACE
- DOX-TACE (Active Comparator): Patients treated by conventional TACE using doxorubicin chemoemulsion
  Interventions: Procedure: DOX-TACE

INTERVENTIONS:
Procedure: IDA-TACE — Stable chemoemulsion will be produced by dissolving 10 mg of idarubicin powder (Zavedos; Pfizer, New York, NY, USA) in 2.5 mL of an iodinated contrast agent. This solution will then be mixed with 10 mL of iodized oil (Lipiodol Ultrafluid; Guerbet, Villepinte, France) using a three-way stopcock. This chemoemulsion will be prepared in aliquots (0.8 mL of chemoemulsion in each 1 mL syringe) and injected until the embolization endpoint is achieved.
  Other Names: Conventional TACE using idarubicin chemoemulsion
  Arms: IDA-TACE
Procedure: DOX-TACE — Stable chemoemulsion will be produced by dissolving 50 mg of doxorubicin powder (Adriamycin RDF; Ildong Pharmaceutical, Seoul, Republic of Korea) in 2.5 mL of an iodinated contrast agent. This solution will then be mixed with 10 mL of iodized oil (Lipiodol Ultrafluid; Guerbet, Villepinte, France) using a three-way stopcock. This chemoemulsion will be prepared in aliquots (0.8 mL of chemoemulsion in each 1 mL syringe) and injected until the embolization endpoint is achieved.
  Other Names: Conventional TACE using doxorubicin chemoemulsion
  Arms: DOX-TACE

SUMMARY:
Little is known about whether the types of chemotherapeutic agents affect the efficacy of transarterial chemoembolization in patients with hepatocellular carcinoma. Although doxorubicin is the most commonly-used chemotherapeutic agent in the world, idarubicin is recently in the spotlight after promising results of the in vitro and prospective single-arm studies. On the other hand, there are many reports showing that the type of chemotherapeutic agents does not significantly alter the efficacy of transarterial chemoembolization. This is a randomized-controlled trial to show the non-inferiority of idarubicin compared to doxorubicin in patients with hepatocellular carcinoma who receive transarterial chemoembolization as the first-line treatment.

DETAILED DESCRIPTION:
Eligible patients will be randomly allocated either in the IDA-cTACE or DOX-cTACE group, and the randomization can be stratified by Child-Pugh class. Each patient will be treated by conventional chemoembolization using a microcatheter and chemoemulsion. For the chemoemulsion preparation method, 10 mg of idarubicin powder (IDA-cTACE) or 50 mg of doxorubicin powder (DOX-cTACE) will be dissolved by 2.5 mL of iodinated contrast media, and then mixed with 10 mL of iodized poppy seed oil (Lipiodol; Lipiodol Ultrafluid, Guerbet, France). The amount of chemoemulsion administered to each patient will be determined by an operator regarding tumor size, vascularity, etc. Additional embolization will be performed using calibrated gelatin sponge particles usually 100-350 µm until the arterial flow is almost stopped. Afterwards, Patients will be evaluated at 1, 3, and 6 months after the initial treatment, but the follow-up can be individualized at the discretion of hepatologists or hepatic surgeons blinded to the treatment allocation. In cases of residual or recurred tumor, additional treatments will be determined by the blinded hepatologists or hepatic surgeons. Once a patient with residual or recurred tumor receives repetitive TACE, the same drug (idarubicin or doxorubicin) used at the initial TACE will be used for re-treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 or above.
2. Patients diagnosed with HCC either histologically and/or radiologically (LI-RADS 4 or 5).
3. Patients with five or fewer tumors.
4. Patients in which the largest tumor is 5 cm or less in diameter.
5. Patients with no prior treatment experience for HCC.
6. Patients categorized as Child-Pugh class A or B.
7. Patients with an Eastern Cooperative Oncology Group performance status of 2 or below.
8. Patients without severe functional abnormalities of major organs: the following results from a blood test conducted within a month prior to the procedure must be satisfied:

   * WBC count ≤ 12,000 / mm3
   * Absolute neutrophil count ≥ 1,500 /mm3
   * Hemoglobin ≥ 8.0 g/dL
   * Total bilirubin ≤ 3.0 mg/dL
   * eGFR ≥ 30 mL/min/1.73 m2
   * Patients deemed clinically most suitable to receive TACE through hepatologist, hepatic surgeon, or multidisciplinary consultation: patients for whom other treatments such as liver transplantation/surgery/ablation are realistically impossible or, even if technically possible, do not have significant clinical benefits compared to TACE.
   * Patients who have understood sufficiently about this clinical trial and have given written consent to participate.
   * Fertile women capable of effective contraception for at least 6.5 months after TACE, and men with fertile female partners capable of effective contraception for at least 3.5 months after TACE.

Exclusion Criteria:

1. Patients with HCC involving the portal vein or hepatic vein.
2. Patients with extrahepatic spread of HCC
3. Patients diagnosed with a cancer other than HCC within 2 years of enrollment.
4. Patients who have undergone a biliary-intestinal anastomosis.
5. Patients for whom the use of idarubicin or doxorubicin is contraindicated (including severe heart failure, arrhythmia, hypersensitivity to anthracycline chemotherapy, pregnant or nursing women, etc.).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-04-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | From the initial TACE to the end of the 6-month follow-up or commencement of subsequent anticancer treatment, whichever comes first
  the number of patients with partial or complete response as the best overall response divided by the total number of participants in the analysis population

SECONDARY OUTCOMES:
3-month tumor response by LI-RADS tumor response criteria | From the initial TACE to the end of the 3-month follow-up or commencement of subsequent anticancer treatment, whichever comes first
3-month tumor response by localized mRECIST | From the initial TACE to the end of the 3-month follow-up or commencement of subsequent anticancer treatment, whichever comes first
3-month tumor response by mRECIST | From the initial TACE to the end of the 3-month follow-up or commencement of subsequent anticancer treatment, whichever comes first
6-month tumor response by LI-RADS tumor response criteria | From the initial TACE to the end of the 6-month follow-up or commencement of subsequent anticancer treatment, whichever comes first
6-month tumor response by localized mRECIST | From the initial TACE to the end of the 6-month follow-up or commencement of subsequent anticancer treatment, whichever comes first
6-month tumor response by mRECIST | From the initial TACE to the end of the 6-month follow-up or commencement of subsequent anticancer treatment, whichever comes first
Time-to-progression | From the date of randomization to tumor progression or study termination (6 months after the last patient is treated), whichever comes first
  Time interval between the first TACE to tumor progression by mRECIST
Adverse event | 30 days
  Common Terminology Criteria for Adverse Events v5.0
Treatment-related serious adverse event | 30 days
  Common Terminology Criteria for Adverse Events v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jin Woo Choi, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi JW, Kim HC, Han J, Jang MJ, Chung JW. Transarterial Chemoembolization Using Idarubicin Versus Doxorubicin Chemoemulsion in Patients with Hepatocellular Carcinoma (IDADOX): Protocol for a Randomized, Non-inferiority, Double-Blind Trial. Cardiovasc Intervent Radiol. 2024 Mar;47(3):372-378. doi: 10.1007/s00270-023-03621-9. Epub 2023 Dec 26. PMID 38147153